CLINICAL TRIAL: NCT04275648
Title: Evaluation of Exercise Induced Bronchoconstriction by Field Test Using Lung Function and a Novel Automated Digital Clinical Decision System
Brief Title: Exercise Induced Bronchoconstriction and Field Tests
Acronym: EXCIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Olympiatoppen, The Norwegian Olympic Sports Centre, Oslo, Norway (Unknown); Norwegian School of Sport Sciences (Other)
Responsible Party: Principal Investigator, Björn Nordlund, PhD, Karolinska Institutet
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: V.4
Record Dates: First submitted 2020-01-27; First posted 2020-02-19 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2022-06

CONDITIONS: Exercise Induced Bronchoconstriction; Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Asthmatuner field tests vs laboratory tests (Experimental): Each participant will perform two standardized field tests either before or after Eucapnic Voluntary Hyperpnea or Methacholine bronchial provocation test. In addition, unstandardized field tests will be performed in case of exercise induced respiratory symptoms.
  Interventions: Diagnostic Test: AsthmaTuner exercise field test

INTERVENTIONS:
Diagnostic Test: AsthmaTuner exercise field test — AsthmaTuner consist of a a bluetooth spirometer and smartphone app with protocol for measuring lung function (FEV1) and perform 8 min exercise challenge test and a healthcare web interface.
  Other Names: AsthmaTuner

SUMMARY:
Asthma and exercise induced bronchoconstriction (EIB) represent an important challenge for the athlete, and correct diagnosis is important as it affects health as well as performance with strict regulations concerning asthma medication. The primary objective of this study on elite athletes with symptoms of EIB, is to assess if EIB can be determined equally by repeated standardized and unstandardized field ECT using AsthmaTuner, and eucapnic voluntary hypernoea (EVH).

Methods: The study has an open design including elite athletes with symptoms of EIB. They will be equipped with an AsthmaTuner to perform 3-5 repeated exercise tests with AsthmaTuner in their natural training and competing environment, followed by an EVH test within four weeks after the first visit. Olympiatoppen is a national clinic in Oslo, Norway, providing health care and screening of elite athletes. At least 60 elite athletes aged 16 to 50 years with a history of EIB symptoms within the last 8 weeks will be invited to participate. The eucapnic voluntarily hyperventilation (EVH) test and two standardized field exercise test will be performed according to guidelines. In addition, the participants will be encouraged to perform unstandardized lung function tests in relation to perceived respiratory symptoms during exercise.

DETAILED DESCRIPTION:
Asthma is the most common chronic condition in Olympic athletes. Asthma is defined as a chronic inflammation in the airways associated with bronchial hyper responsiveness (BHR). It is suggested that there are two phenotypes of asthma among athletes; the classic asthma with early childhood onset and allergic sensitization, and the "sports asthma". While exercise-induced "sports" asthma (EIA) describes symptoms and signs of asthma provoked by exercise, exercise-induced bronchoconstriction (EIB) is defined as the transient narrowing of the lower airway after exercise. In the general population, EIB with or without asthma affects 5% to 20%, but the rate is estimated to be even higher in top athletes participating in winter and summer endurance sports.

Asthma and EIB represent an important challenge for the athlete, and correct diagnosis is important as it affects health as well as performance with strict regulations concerning asthma medication. A clear diagnosis of asthma with confirmation of BHR is strongly suggested by the International Olympic Committee (IOC) and the World Anti-Doping Agency (WADA) before the use of anti-asthmatic medication.

Presence of BHR is demonstrated by direct or indirect bronchial provocation testing. Direct bronchial provocation causes bronchoconstriction by acting on specific airway receptors on the bronchial smooth muscle, while indirect bronchial provocation tests acts indirectly via the release of contractile mediators. Direct bronchial provocation via inhalation of methcacholine has been reported to be highly sensitive in detecting BHR in elite athletes, and is the method of choice at Olympiatoppen, Norway. To reduce the risk of false positive BHR results, methacholine provocation is only used in patients with symptoms of EIA. Less sensitive but more specific, is indirect bronchial provocation including several methods for the diagnosis of EIB. The most intuitive is exercise (field and laboratory) challenge testing (ECT), but sensitivity has been reported to be low, since exercise load and intensity have large impact on ability to detect EIB and in field-testing (FT), standardizing ambient conditions are impossible. By eucapnic voluntary hyperpnoea (EVH) of dry air, the two components of EIB are induced: The inflammatory cascade in the airways causing airway smooth muscle contraction, and airway oedema. The EVH has been endorsed by the IOC-MC as the gold standard due to its high specificity, but for mild to moderate EIB, EVH has wide sensitivity, specificity and poor repeatability, which may rely on inability to simulate the competition environment. Suboptimal tests for EIB may explain why previous papers report poor relationship between symptoms of EIA and the objective EIB in athletes, leaving the actual rate of EIB remains unclear. What has been argued to be the true "gold standard" is a sports-specific exercise FT , performed in the actual training conditions which also makes it easier for the athlete to perform at maximum exercise. The advantages of monitoring with peak expiratory flow (PEF) or forced expiratory volume in 1 s (FEV1) outside a laboratory with a PEF meter or spirometer, respectively, are that it is simple and cheap. It also enables measure of bronchial challenge testing in close relationship to symptoms, since laboratory bronchial challenge testing often are negative in subjects being away from their profession too long. Due to lack of standardization, it is recommended to measure serial lung function after a specific exercise in at least two different time-points. However, traditional non-digital method of serial PEF/FEV1 monitoring has limitations with poor adherence, interpretation difficulties with objectivity and time-consuming analysis and reading of paper PEF/FEV1 plots.

Recently, AsthmaTuner (Medituner AB) consisting of a patient smartphone application, a portable wireless spirometer for measuring lung function (PEF/FEV1), and a healthcare interface including treatment plan, was reported to significantly improve management of uncontrolled asthma. Such electronically clinical decision support systems (CDSS) has gained acceptance for the diagnosis of asthma, and by the ability to assess patient generated data in field ECTs, the CE-marked AsthmaTuner may provide athletes a feasible, time and cost-efficient self-monitoring of EIB and asthma. AsthmaTuner may also empower athletes in monitoring their lung function over time. These lung function measurements contain unexpected amounts of information for identifying athletes with distinct phenotypes of EIB due to strenuous sports and environmental conditions. Hence, AsthmaTuner have the potential to fill the knowledge gap regarding prevalence of EIB, development of EIB and the lack of association between symptoms and detection of EIB in athletes.

Objective and aims The primary objective of this study on elite athletes with symptoms of EIB, is to assess if EIB can be determined equally by repeated standardized and unstandardized field ECT using AsthmaTuner, and EVH.

Specific research aims include:

1. The primary aim is to identify the prevalence of EIB using AsthmaTuner in repeated field ECT.
2. The secondary aim is to investigate the reproducibility of AsthmaTuner.
3. The third aim is to compare EIB detected by repeated field ECT using AsthmaTuner with standardized EVH.
4. The fourth aim is to compare BHR defined by methacholine bronchial provocation test, field testing and EVH.

Material and Methods Design The study has an open design including elite athletes with symptoms of EIB. They will be equipped with an AsthmaTuner to perform 3-5 repeated exercise tests with AsthmaTuner in their natural training and competing environment, followed by an EVH test within four weeks after the first visit.

Study population Olympiatoppen is a national clinic in Oslo, Norway, providing health care and screening of elite athletes. At least 60 elite athletes aged 16 to 50 years with a history of EIB symptoms within the last 8 weeks and ability to comply with the study protocol will be invited to participate. The athletes will be recruited before or after clinical visits with laboratory testing of EIB at Olympiatoppen, as well as eligible students at Norwegian School of Sport Sciences. the National Patients who enter the study, will not start or receive additional asthma treatment until completion of the study. If already on asthma treatment, beta2-agonists and triatropiumpromide will be stopped prior to methacholine bronchial provocation, standardized and unstandardized exercise FT and EVH, according to the guidelines.

Eucapnic voluntarily hyperventilation The eucapnic voluntarily hyperventilation (EVH) test will be performed according to guidelines. A single-stage protocol will be used that requires participants to maintain a minute ventilation (VE) close to 85 % of their maximal voluntary ventilation (MVV) for 6 min. During the test, the participants will breathe through a mouthpiece and inspire a gas mixture of 21 % oxygen, 5 % carbon dioxide, with a balance of nitrogen to achieve this target ventilation and simultaneously maintain eucapnia (perform hyperpnea). The inspired gas is administered from two gas cylinders via a commercial system (EucapSys SMTEC, Switzerland). Maximal flow volume loops will be recorded at baseline and 1-20 minutes after the challenge according to international guidelines for standardization of spirometry. The test is considered to be highly sensitive for asthma and is deemed positive if the FEV1 falls ≥10 % from the baseline measurement within 20 min of challenge cessation.

Participants using asthma medications will be specifically instructed to not use their medications prior to the test. All participants will be instructed to avoid strenuous exercise, heavy meals, caffeine containing food or beverage and nicotine 4 h before the test.

Field exercise test with AsthmaTuner The field exercise test will be performed according to guidelines for the diagnosis of EIB (19, 25). A heart rate of 85% of max value during 8 minutes is demanded throughout the exercise test. The subjects need to refrain physical activity and use of short- and long-acting beta-2 agonists and ipratropriumbromide 12 prior to the challenge. All tests are separated by at least 24 hours and performed between 8:30 am and 12 pm to control for diurnal variation in airway caliber. A fall in FEV1 >10% conducted 1, 5, 10, 15, 30 min after exercise confirm current EIB. In addition, the participants will be encouraged to perform unstandardized lung function tests in relation to perceived respiratory symptoms during exercise. Possible fall in FEV1 will be calculated in relation to previously established baseline measurements of FEV1.

Questionnaires Athletes will fill in a structured electronic questionnaire sent by mail concerning demographic background factors, respiratory health, treatment, and healthcare utilization at study enrolment and answer questions about usability and feasibility of using AsthmaTuner at study end.

Statistical analyses The statistical power analysis is based upon the data provided by Rundell et al., reporting that the mean of the pairwise differences between FT and EVH is 0.014 percentage points, with a standard deviation of 8.35 percentage points. Including a drop out rate of 10%, including 60 athletes would provide a power of 80% at a five percent significance level.

Receiver-operating characteristic (ROC) curve will be plotted for EVH with Spearmen's rank correlations to estimate the predictive values of the exercise test maximal fall in PEF/FEV1 with AsthmaTuner. The optimal cut-off level for sensitivity and specificity will be estimated based on the area under the curve of EVH and FT by AsthmaTuner. Evaluation of the repeatability of AsthmaTuner will be analysed by plotting against the mean of two measurements.

ELIGIBILITY:
Inclusion Criteria:

* History of EIB symptoms within the last 8 weeks will be invited to participate

Exclusion Criteria:

* Additional asthma treatment until completion of the study.
* Athletes will be excluded if any of following criterion is fulfilled; FEV1 <75%, a forced vital capacity <80%, a recent course of oral corticosteroids or infections, as well as pregnancy, chronic diseases or inability to perform the study procedures.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Standardized field exercise test | Change from baseline FEV1 by 30 minutes post exercise
  Forced expiratory volume of one second (FEV1), given by the AsthmaTuner

SECONDARY OUTCOMES:
Unstandardised field exercise test | Change from baseline FEV1 by 30 minutes post exercise
  Forced expiratory volume of one second (FEV1), given by the AsthmaTuner compared with baseline FEV1
EVH | Change from baseline FEV1 by 20 minutes post EVH challenge
  Forced expiratory volume of one second (FEV1) post challenge
Bronchial hyperresponsiveness | Change from baseline FEV1 at 1 minute of last dose given 20% reduction of FEV1 according to the standardised protocol
  <4 µmol cumulated methacholine given to achieve a 20% reduction of FEV1

CONTACTS AND LOCATIONS:
Overall Officials: Björn Nordlund, PhD, Principal Investigator — Women's and Children's Health, Karolinska Institutet
Locations (1):
- Olympiatoppen, Oslo, Norway

REFERENCES:
- [Background] Fitch KD. An overview of asthma and airway hyper-responsiveness in Olympic athletes. Br J Sports Med. 2012 May;46(6):413-6. doi: 10.1136/bjsports-2011-090814. Epub 2012 Jan 8. PMID 22228581
- [Background] Couto M, Stang J, Horta L, Stensrud T, Severo M, Mowinckel P, Silva D, Delgado L, Moreira A, Carlsen KH. Two distinct phenotypes of asthma in elite athletes identified by latent class analysis. J Asthma. 2015;52(9):897-904. doi: 10.3109/02770903.2015.1067321. Epub 2015 Sep 17. PMID 26377281
- [Background] Carlsen KH, Anderson SD, Bjermer L, Bonini S, Brusasco V, Canonica W, Cummiskey J, Delgado L, Del Giacco SR, Drobnic F, Haahtela T, Larsson K, Palange P, Popov T, van Cauwenberge P; European Respiratory Society; European Academy of Allergy and Clinical Immunology. Exercise-induced asthma, respiratory and allergic disorders in elite athletes: epidemiology, mechanisms and diagnosis: part I of the report from the Joint Task Force of the European Respiratory Society (ERS) and the European Academy of Allergy and Clinical Immunology (EAACI) in cooperation with GA2LEN. Allergy. 2008 Apr;63(4):387-403. doi: 10.1111/j.1398-9995.2008.01662.x. PMID 18315727
- [Background] Weiler JM, Bonini S, Coifman R, Craig T, Delgado L, Capao-Filipe M, Passali D, Randolph C, Storms W; Ad Hoc Committee of Sports Medicine Committee of American Academy of Allergy, Asthma & Immunology. American Academy of Allergy, Asthma & Immunology Work Group report: exercise-induced asthma. J Allergy Clin Immunol. 2007 Jun;119(6):1349-58. doi: 10.1016/j.jaci.2007.02.041. Epub 2007 Apr 16. No abstract available. PMID 17433829
- [Background] Norqvist J, Eriksson L, Soderstrom L, Lindberg A, Stenfors N. Self-reported physician-diagnosed asthma among Swedish adolescent, adult and former elite endurance athletes. J Asthma. 2015;52(10):1046-53. doi: 10.3109/02770903.2015.1038389. Epub 2015 Aug 18. PMID 26288032
- [Background] Larsson K, Ohlsen P, Larsson L, Malmberg P, Rydstrom PO, Ulriksen H. High prevalence of asthma in cross country skiers. BMJ. 1993 Nov 20;307(6915):1326-9. doi: 10.1136/bmj.307.6915.1326. PMID 8257888
- [Background] Price OJ, Ansley L, Menzies-Gow A, Cullinan P, Hull JH. Airway dysfunction in elite athletes--an occupational lung disease? Allergy. 2013 Nov;68(11):1343-52. doi: 10.1111/all.12265. Epub 2013 Oct 11. PMID 24117544
- [Background] Brannan JD, Koskela H, Anderson SD. Monitoring asthma therapy using indirect bronchial provocation tests. Clin Respir J. 2007 Jul;1(1):3-15. doi: 10.1111/j.1752-699X.2007.00004.x. PMID 20298272
- [Background] Anderson SD, Kippelen P. Airway injury as a mechanism for exercise-induced bronchoconstriction in elite athletes. J Allergy Clin Immunol. 2008 Aug;122(2):225-35; quiz 236-7. doi: 10.1016/j.jaci.2008.05.001. Epub 2008 Jun 12. PMID 18554705
- [Background] Langdeau JB, Turcotte H, Desagne P, Jobin J, Boulet LP. Influence of sympatho-vagal balance on airway responsiveness in athletes. Eur J Appl Physiol. 2000 Nov;83(4 -5):370-5. doi: 10.1007/s004210000306. PMID 11138577
- [Background] Hull JH, Ansley L, Price OJ, Dickinson JW, Bonini M. Eucapnic Voluntary Hyperpnea: Gold Standard for Diagnosing Exercise-Induced Bronchoconstriction in Athletes? Sports Med. 2016 Aug;46(8):1083-93. doi: 10.1007/s40279-016-0491-3. PMID 27007599
- [Background] Rundell KW, Anderson SD, Spiering BA, Judelson DA. Field exercise vs laboratory eucapnic voluntary hyperventilation to identify airway hyperresponsiveness in elite cold weather athletes. Chest. 2004 Mar;125(3):909-15. doi: 10.1378/chest.125.3.909. PMID 15006949
- [Background] Carlsen KH, Engh G, Mork M. Exercise-induced bronchoconstriction depends on exercise load. Respir Med. 2000 Aug;94(8):750-5. doi: 10.1053/rmed.2000.0809. PMID 10955749
- [Background] Anderson SD. How does exercise cause asthma attacks? Curr Opin Allergy Clin Immunol. 2006 Feb;6(1):37-42. doi: 10.1097/01.all.0000199797.02423.78. PMID 16505610
- [Background] Anderson SD, Argyros GJ, Magnussen H, Holzer K. Provocation by eucapnic voluntary hyperpnoea to identify exercise induced bronchoconstriction. Br J Sports Med. 2001 Oct;35(5):344-7. doi: 10.1136/bjsm.35.5.344. PMID 11579071
- [Background] Ansley L, Kippelen P, Dickinson J, Hull JH. Misdiagnosis of exercise-induced bronchoconstriction in professional soccer players. Allergy. 2012 Mar;67(3):390-5. doi: 10.1111/j.1398-9995.2011.02762.x. Epub 2011 Dec 17. PMID 22175650
- [Background] Rundell KW, Im J, Mayers LB, Wilber RL, Szmedra L, Schmitz HR. Self-reported symptoms and exercise-induced asthma in the elite athlete. Med Sci Sports Exerc. 2001 Feb;33(2):208-13. doi: 10.1097/00005768-200102000-00006. PMID 11224807
- [Background] Heir T, Larsen S. The influence of training intensity, airway infections and environmental conditions on seasonal variations in bronchial responsiveness in cross-country skiers. Scand J Med Sci Sports. 1995 Jun;5(3):152-9. doi: 10.1111/j.1600-0838.1995.tb00029.x. PMID 7552758
- [Background] Parsons JP, Hallstrand TS, Mastronarde JG, Kaminsky DA, Rundell KW, Hull JH, Storms WW, Weiler JM, Cheek FM, Wilson KC, Anderson SD; American Thoracic Society Subcommittee on Exercise-induced Bronchoconstriction. An official American Thoracic Society clinical practice guideline: exercise-induced bronchoconstriction. Am J Respir Crit Care Med. 2013 May 1;187(9):1016-27. doi: 10.1164/rccm.201303-0437ST. PMID 23634861
- [Background] Ljungberg H, Carleborg A, Gerber H, Ofverstrom C, Wolodarski J, Menshi F, Engdahl M, Eduards M, Nordlund B. Clinical effect on uncontrolled asthma using a novel digital automated self-management solution: a physician-blinded randomised controlled crossover trial. Eur Respir J. 2019 Nov 14;54(5):1900983. doi: 10.1183/13993003.00983-2019. Print 2019 Nov. PMID 31481605
- [Background] Matui P, Wyatt JC, Pinnock H, Sheikh A, McLean S. Computer decision support systems for asthma: a systematic review. NPJ Prim Care Respir Med. 2014 May 20;24:14005. doi: 10.1038/npjpcrm.2014.5. PMID 24841952
- [Background] Courbis AL, Murray RB, Arnavielhe S, Caimmi D, Bedbrook A, Van Eerd M, De Vries G, Dray G, Agache I, Morais-Almeida M, Bachert C, Bergmann KC, Bosnic-Anticevich S, Brozek J, Bucca C, Camargos P, Canonica GW, Carr W, Casale T, Fonseca JA, Haahtela T, Kalayci O, Klimek L, Kuna P, Kvedariene V, Larenas Linnemann D, Lieberman P, Mullol J, Ohehir R, Papadopoulos N, Price D, Ryan D, Samolinski B, Simons FE, Tomazic P, Triggiani M, Valiulis A, Valovirta E, Wagenmann M, Wickman M, Yorgancioglu A, Bousquet J. Electronic Clinical Decision Support System for allergic rhinitis management: MASK e-CDSS. Clin Exp Allergy. 2018 Dec;48(12):1640-1653. doi: 10.1111/cea.13230. Epub 2018 Aug 20. PMID 29999223
- [Background] Frey U, Brodbeck T, Majumdar A, Taylor DR, Town GI, Silverman M, Suki B. Risk of severe asthma episodes predicted from fluctuation analysis of airway function. Nature. 2005 Dec 1;438(7068):667-70. doi: 10.1038/nature04176. PMID 16319891
- [Derived] Reier-Nilsen T, Stang JS, Flatsetoy H, Isachsen M, Ljungberg H, Bahr R, Nordlund B. Unsupervised field-based exercise challenge tests to support the detection of exercise-induced lower airway dysfunction in athletes. BMJ Open Sport Exerc Med. 2023 Jul 24;9(3):e001680. doi: 10.1136/bmjsem-2023-001680. eCollection 2023. PMID 37520311